CLINICAL TRIAL: NCT06860230
Title: Evaluation of NellcorTM Pulse Oximetry Accuracy With the Philips picoSAT X SpO2 Board With Fourier Artifact Suppression Technology in Adult Volunteers
Brief Title: Philips FAST Evaluation
Acronym: NELFST
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Collaborators: Philips Medical Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT24049NELFST
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-01

CONDITIONS: Oxygen Saturation Measurement
Keywords: pulse oximetry; Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Healthy Volunteers: All subjects who meet the inclusion criteria are enrolled into the test group and participate in data collection have the Philips FAST SpO2 with Nellcor Pulse Oximetry Sensors
  Interventions: Device: Philips FAST SpO2 with Nellcor Pulse Oximetry Sensors

INTERVENTIONS:
Device: Philips FAST SpO2 with Nellcor Pulse Oximetry Sensors — Noninvasive pulse oximeter

SUMMARY:
Evaluation of Philips FAST technology with Nellcor sensors

DETAILED DESCRIPTION:
Evaluate saturation accuracy claims for the Philips picoSAT X SpO2 board with FAST algorithm, paired with Nellcor™ sensors in a diverse subject population, over a specified saturation range

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 and < 51 years of age
2. Subject is willing and able to comply with study procedures and duration
3. Subject is willing to sign an informed consent
4. Subject weighs >40kg
5. Subject is a non-smoker or has not smoked within 36 hours prior to the study
6. Cleared same day health assessment form and health screening

Exclusion Criteria:

1. Subject is considered as being morbidly obese (defined as BMI >39.5)
2. Compromised circulation, injury, or physical malformation of fingers, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the sites utilized)
3. Participants of childbearing potential who are pregnant, who are trying to get pregnant, or who have a urine test positive for pregnancy on the day of the study
4. Subjects with COHb levels >3% as assessed by CO-Oximetry during the procedure
5. tHb < 10 g/dl as assessed by CO-Oximetry during the procedure
6. MetHb ≥ 2% as assessed by CO-Oximetry during the procedure
7. Subjects with known respiratory conditions such as:

   1. uncontrolled / severe asthma
   2. flu or influenza type infection
   3. pneumonia / bronchitis
   4. shortness of breath / respiratory distress
   5. unresolved respiratory or lung surgery
   6. emphysema, COPD, lung disease
   7. recent COVID (last 2 months)
8. Subjects with known heart or cardiovascular conditions such as:

   1. hypertension: systolic pressure >140mmHg, or diastolic pressure >90mmHg on 3 consecutive readings
   2. previous cardiovascular surgery
   3. chest pain (angina)
   4. heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
   5. previous heart attack
   6. blocked artery
   7. unexplained shortness of breath
   8. congestive heart failure (CHF)
   9. history of stroke
   10. transient ischemic attack
   11. carotid artery disease
   12. myocardial ischemia
   13. myocardial infarction
   14. cardiomyopathy
   15. implantable active medical device such as pacemaker or automatic defibrillator
9. Self-reported health conditions as identified in the Health Assessment Form

   1. diabetes
   2. uncontrolled thyroid disease
   3. kidney disease / chronic renal impairment
   4. history of seizures (except childhood febrile seizures)
   5. epilepsy
   6. history of unexplained syncope
   7. recent history of frequent migraine headaches
   8. recent symptomatic head injury, within the last 2 months
   9. cancer requiring chemotherapy, radiation, or current treatment
   10. subjects with known clotting disorders
   11. history of bleeding disorders or personal history of prolonged bleeding from injury
   12. history of blood clots
   13. hemophilia
   14. sickle cell trait or disease
   15. current use of blood thinner: prescription or daily use of aspirin
   16. subjects with Severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors
   17. participants with severe allergy to iodine (only applicable if iodine is used)
   18. subjects with prior or known severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocain) or heparin
   19. arterial cannulation within the last 30 days prior to study date, (this may exclude only one radial artery site, left or right)
   20. history of clinically significant complications from previous arterial cannulation
   21. Failure of Allen's test
   22. unwillingness or inability to remove colored nail polish or colored artificial nails other than clear from test digits
   23. other known health condition, upon disclosure in Health Assessment form at PI's discretion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects ≥ 18 and < 51 years of age, with varying skin tones and diversity across ethnicity, race, gender, and sex assigned at birth.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of Saturation Accuracy | 2 - 3 hours
  Performance will be determined by calculating the accuracy in terms of root mean square difference (ARMS) comparing the noninvasive oxygen saturation measurement (SpO2) to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Randall M Clark, M.D., Principal Investigator — Medtronic Clinical Physiology Lab
Locations (1):
- Medtronic Clinical Physiology Lab, Denver, Colorado, United States